CLINICAL TRIAL: NCT07243990
Title: The Effect of Neuromonitoring on the Incidence of Postoperative Agitation in Pediatric Patients Undergoing General Anesthesia
Brief Title: Impact of Neuromonitoring on Postoperative Agitation in Pediatric General Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Esin Topkara Oğur, MD, Anesthesiology Specialist, Sakarya University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-SEAH-ETO-DSA
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Agitation; Emergence Delirium, Anesthesia
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Monitoring-Based Care (Experimental): After the patients are taken into the operating room, they will be monitored. This monitoring will include tracking brain activity using DSA (Depth of Sedation Assessment), and anesthesia induction will be performed under this monitoring.
  Interventions: Device: dsa intervention group
- Group Standart Care (Experimental): After the patients are taken into the operating room, they will be monitored, and anesthesia induction will be performed using the traditional method by administering anesthetic agents based on body weight.
  Interventions: Other: Traditional Monitoring

INTERVENTIONS:
Device: dsa intervention group — The Density Spectral Array (DSA) device, developed for use in operating rooms, facilitates the interpretation of Electroencephalogram (EEG) data and guides the anesthesiologist. In our operating room, patients under anesthesia are also monitored using this device.
  Arms: Group Monitoring-Based Care
Other: Traditional Monitoring — This group will receive anesthesia induction using the traditional method, and monitoring will continue simultaneously with EEG (Electroencephalography).
  Arms: Group Standart Care

SUMMARY:
Postoperative agitation is frequently observed in the pediatric patient group following general anesthesia. The exact cause of this agitation has not been clearly determined; however, it may be associated with various factors such as anesthesia depth, family approach, postoperative pain, or unpleasant odors perceived by the child. The depth of anesthesia is indirectly monitored by observing the patient's blood pressure, heart rate, and oxygen saturation, as well as by assessing the alveolar concentration of the inhalation agent. Patients under anesthesia are in a state of deep sleep. In recent years, this sleep state has begun to be monitored more closely with the development of new devices.

Electroencephalography (EEG) is a test that records and measures the brain's electrical activity, providing information about the depth of sleep according to the patient's brain activity. The Density Spectral Array (DSA) device, developed for use in operating rooms, facilitates the interpretation of EEG data and guides the anesthesiologist. In our operating room, patients under anesthesia are also monitored using this device.

Our aim is to evaluate emergence agitation in patients monitored with this device compared to those who are not monitored.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 6-12 years

Without chronic comorbid conditions

No history of epilepsy

Presenting for surgery with preserved consciousness, oriented and cooperative

Exclusion Criteria:

Intracranial surgeries

Intellectual disability

Emergency trauma cases

Forehead area unsuitable for electrode placement

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative agitation after postoperative 30 minutes | First 30 minutes in the postoperative care unit after emergence from anesthesia.
  Richmond Agitation-Sedation Scale (RASS) (-5 to +4) will be recorded at 0, 5, 10, 15, and 30 minutes after emergence in the postoeperative care unit. For each participant, the highest (maximum) RASS value observed within the first 30 minutes will be analyzed as the primary outcome. Higher scores indicate more severe agitation. The Richmond Agitation-Sedation Scale (RASS) is used to assess a patient's level of agitation or sedation. Scores range from +4 to -5, where +4 represents the most severe agitation and -5 represents unarousable sedation. Higher positive scores indicate more severe agitation, while lower negative scores indicate deeper sedation.